CLINICAL TRIAL: NCT00102219
Title: A Phase 2 Study of ALIMTA Plus Doxorubicin Administered Every 21 Days in Patients With Advanced Breast Cancer
Brief Title: A Study of Pemetrexed Plus Doxorubicin Given to Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8426; H3E-MC-JMGV
Record Dates: First submitted 2005-01-25; First posted 2005-01-26 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Pemetrexed; Doxorubicin

INTERVENTIONS:
Drug: Pemetrexed
Drug: Doxorubicin

SUMMARY:
This is a non-randomized Phase 2 study testing pemetrexed and doxorubicin in combination for locally advanced or metastatic breast cancer. Both pemetrexed and doxorubicin have been combined with other drugs, but they have not yet been combined with each other. It is expected that the patient will benefit from the different mechanisms of action of the two drugs. However, there is no guarantee that the patient will benefit from this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic breast cancer that is not amenable to local treatment.
* Patients must be chemo-naive or have received only neoadjuvant and/or adjuvant chemotherapy.
* At least one measurable lesion.
* No chemotherapy within 4 weeks prior to enrollment.
* Signed informed consent from the patient.

Exclusion Criteria:

* Prior chemotherapy for metastatic breast cancer.
* Prior treatment with any anthracyclines or anthracenedione-containing regimen.
* Treatment within the last 30 days with any drug that has not received regulatory approval.
* Pregnancy and/or breast feeding.
* Inability or unwillingness to take folic acid or vitamin B12 supplementation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2004-10; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To assess the antitumor activity of pemetrexed plus doxorubicin, as measured by overall tumor response rate

SECONDARY OUTCOMES:
Time to progressive disease
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Belo Horizonte, BH
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, São Paulo, São Paulo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rio de Janeiro
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Athens, Greece
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Székesfehérvár
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lima, Peru
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lodz
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Valencia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Caracas, Venezuela

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com